CLINICAL TRIAL: NCT04715984
Title: Corticostriatal Neurophysiology in Parkinson's Disease Cognitive Impairment
Brief Title: Corticostriatal Contributions to Parkinson's Disease Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Bick, Assistant Professor of Neurosurgery, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201868
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neural recordings and stimulation (Experimental)
  Interventions: Other: Neurophysiology recordings; Other: Neural stimulation

INTERVENTIONS:
Other: Neurophysiology recordings — Neurophysiology recordings will be performed during deep brain stimulation surgery and their relationship to performance on a gambling task evaluated
Other: Neural stimulation — Neural stimulation will be delivered during a gambling task and its impact on task performance quantified

SUMMARY:
The goal of this study is to learn more about the brain activity underlying Parkinson's disease cognitive impairment. The investigators will utilize neural recordings from corticostriatal structures performed during deep brain stimulation surgery to measure neural activity underlying nonmotor symptoms of Parkinson's disease.

ELIGIBILITY:
Inclusion criteria:

* Scheduled to undergo deep brain stimulation surgery under local anesthesia at Vanderbilt University Medical Center
* Planned clinical electrode trajectory that contacts caudate
* Age greater than or equal to 40
* Diagnosis of Parkinson's disease
* Able to participate in intraoperative testing
* English speaking

Exclusion criteria:

* Age less than 40
* Not able to participate in intraoperative testing (for example unable to comprehend instructions or follow directions)
* Movement disorder other than Parkinson's disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Changes in caudate DLPFC beta coherence | Baseline to end of Deep Brain Stimulation (DBS), approximately 3-4 hours
  Caudate DLPFC coherence will be computed at rest and during the gambling task and correlated with cognitive metrics
Changes in gambling task performance with neural stimulation | Baseline to end of Deep Brain Stimulation (DBS), approximately 3-4 hours
  The gambling task will involve seeing a series of cards presented on the screen and pressing a button to respond with a bet. Gambling task performance will be compared between stimulated and non stimulated blocks and between stimulation targets

SECONDARY OUTCOMES:
Change in beta power with neural stimulation | Baseline to end of deep brain stimulation (DBS) surgery, approximately 3-4 hours
  Beta power will be computed and compared between stimulation on and off conditions for different targets

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bick, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No